

## INFORMED CONSENT INFORMATION DOCUMENT

Improving the Quality of Smoking Cessation and Shared Decision Making for Lung Cancer Screening: A Cluster Randomized Trial 2019-0265

Subtitle: Patient Baseline Questionnaire Statement

Study Chair: Robert Volk

The goal of this research study is to find the best ways to help people quit smoking and make informed decisions about lung cancer screening. If you agree to take part in this study, your primary care provider or a Quitline counselor will speak to you about lung cancer screening and quitting smoking.

If you are in group 1, you will talk with your primary care provider at your upcoming visit about lung cancer screening and smoking cessation. If you are in group 2, you will receive up to 6 smoking cessation counseling sessions over the phone to help you quit smoking and to teach you about lung cancer screening. The first session will take place before your upcoming appointment with your primary care provider.

You will be asked some research questions at four different times: at the start of the study (you may complete those now) and at follow-ups 1 week, 8 weeks, and 12 weeks after your upcoming primary care visit.

You will be mailed a reloadable gift card to compensate you for your time and effort to complete the research visits. The card will be loaded with \$25 after you complete the 1-week visit (V1), \$25 after you complete the 8-week visit (V2), and with \$40 after you complete the 12-week visit (V3). You will receive an extra \$10 for each visit questionnaire you complete early, for a total of up to \$130. You will not receive partial payment for incomplete visits, and you will not be compensated for counseling calls.

Questionnaires will be considered completed early if you submit them within 5 days of receiving the link.

You will speak with an MD Anderson study staff member during your upcoming phone visit and more details of the study will be discussed with you. You will be asked for your consent to participate in the study at that time. In preparation for your phone visit, you may complete the attached questionnaires, which will help lower the amount of time needed to complete the phone visit. Additional information about the study is also

attached and will be discussed with you in more detail during the phone visit. If you complete the questions but choose not to participate in the full study, your data will be kept.

The questionnaires attached will ask you about smoking behavior and alcohol use, health and mental health history, emotions, motivation, withdrawal symptoms, decision making, risks of smoking, knowledge about lung cancer screening, and quality of life. These questionnaires should take about 40 to 50 minutes total to complete.

## **Questionnaire Statement**

I have read the description of the study, and I have decided to answer the questionnaires attached and described here. I understand that I may refuse to answer any (or all) of the questions at this time and I am free to refuse study participation if I wish.

During the course of this study, the research team at The University of Texas MD Anderson Cancer Center (MD Anderson) will be collecting information about me that they may share with health authorities, study monitors who check the accuracy of the information, and individuals who put all the study information together in report form. By answering the questions, I am providing authorization for the research team to use and share my information at any time. If I do not want to authorize the use and disclosure of my information, I may choose not to answer these questions. There is no expiration date for the use of this information as stated in this authorization.

I may withdraw my authorization at any time, in writing, for any reason as long as that information can be connected to me. I can learn more about how to withdraw my authorization by calling the Chair of MD Anderson's IRB at 713-792-6477 or by contacting the study chair, Dr. Robert Volk at 713-563-0020.

\_\_\_\_\_

**Questionnaires Link**